CLINICAL TRIAL: NCT00269100
Title: Prevention of Bacteremia Induced by Debridement of Pressure Ulcer
Status: Terminated | Type: Observational
Sponsor: Herzog Hospital (Other)
Other Study IDs: Jaul1CTIL
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Pressure Ulcers; Bacteremia
Keywords: Debridement
MeSH Terms: conditions — Pressure Ulcer; Bacteremia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to analyse bacteremia induced by debridement of pressure ulcers in patients in the complex nursing department.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the complex nursing department
* With contaminated pressure ulcers
* Going to have a debridement procedure

Exclusion Criteria:

* Penicillin sensitivity
* Bacteremia that does not react to the antibiotic treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Overall Officials: Efraim Jaul, Study Director — Herzog Hospital
Locations (1):
- Herzog Hospital, Jerusalem, Israel